CLINICAL TRIAL: NCT06483750
Title: The Efficacy of the Systane iLux System on Preoperative Cataract Patients on Dry Eye Disease Due to Meibomian Gland Dysfunction
Brief Title: Preoperative iLux on Cataract Surgery Derived Dry Eye Disease Due to Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCR245538
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease; Meibomian Gland Dysfunction; Cataract Senile; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control: No Systane iLux Treatment (No Intervention): No Systane iLux treatment at baseline visit two weeks prior to cataract surgery.
- Systane iLux Treatment (Experimental): Systane iLux administration at baseline visit two weeks prior to cataract surgery.
  Interventions: Device: Systane iLux Treatment

INTERVENTIONS:
Device: Systane iLux Treatment — The Systane iLux is an approved thermal pulsation device to treat dry eye disease. The application of heat and compression to both eyelids melts meibum in the obstructed glands to restore the secretion and production of meibum to the eye. The Systane iLux will only be administered to the eye to undergo cataract surgery.
  Arms: Systane iLux Treatment

SUMMARY:
This prospective study will investigate the effect of pre-operative Systane iLux system administration in treated cataract induced dry eye disease.

DETAILED DESCRIPTION:
Eligible patients to be recruited will have scheduled upcoming senile cataract surgery. Enrolled patients in the active arm (n=25) will receive pre-operative Systane iLux treatment two weeks prior to surgery at the baseline visit. Patients in the control arm will receive no Systane iLux treatment at the baseline visit two weeks prior to cataract surgery. Patients will be assessed on baseline metrics for dry eye disease stemming and meibomian gland dysfunction (MGD) at the baseline visit two weeks prior to cataract surgery. These metrics include tear break up time (TBUT), standard patient evaluation of eye dryness questionnaire (SPEED), ocular surface and surface disease index (OSDI) surveys, and lipid layer thickness (LLT). At the follow up visit four weeks after cataract surgery, these same metrics will be assessed again for any significant changes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 at the time of informed consent
* Must understand; be willing and able, and likely to fully comply with study procedures, visit schedule, and restrictions
* Upcoming scheduled senile cataract surgery

Exclusion Criteria:

* Eyelid abnormalities
* Patients with active ocular infection, active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Ocular surgery within the last 6 months
* Occlusion therapy with lacrimal or punctum plugs within the last 3 months
* Patients with an ocular surface abnormality that may compromise corneal integrity
* Patients with ocular injury or trauma, chemical burns, or limbal stem cell deficiency (within prior 3 months)
* Patients with cicatricial lid margin disease
* patients with lid surface abnormalities that affect lid function in either eye; patients with aphakia
* Patients with permanent makeup or tattoos on their eyelids.
* Previous application/administration of Systane iLux or LipiFlow treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Changed in Lipid Layer Thickness (LLT) measurement from baseline visit | 6 weeks
  To assess improvement in tear film lipid layer by imaging through LipiView II. Thin lipid layer thickness (<60 nm) indicates a tear film instability and therefore an increased evaporation rate, high osmolarity, and dry eye symptoms. In contrast, a thicker lipid layer thickness (<120 nm) indicates a more stable tear film stability

SECONDARY OUTCOMES:
Change in standard patient evaluation of eye dryness questionnaire (SPEED) questionnaire from baseline visit | 6 weeks
  To assess the improvement of dry eye symptoms by SPEED questionnaire. 0 score is the minimum (no dry eye symptom); 64 is the maximum score (most symptomatic). Change = (Follow up visit score - Baseline score)
Mean change from baseline of Fluorescein Tear Break-Up Time (TBUT) from baseline visit | 6 weeks
  The shorter the TBUT, the lower the tear film stability. Lower tear film stability is associated with dry eye. Change = (Follow up visit value - baseline visit value). shorter the TBUT, the lower the tear film stability. Lower tear film stability is associated with dry eye. Change = (Follow up visit value - baseline visit value).
Change in ocular surface and disease index (OSDI) score questionnaire from baseline visit | 6 weeks
  The OSDI survey provides a score from 0 to 100 with a higher score indicating a more severe symptoms of dry eye disease. A normal score fro patients without dry eye would be 12 or below, while a score of 13 to 22 indicates mild disease, 23 to 32 indicates moderate disease, and patients with a score above 33 are characterized as having severe eye disease. Change = (Follow up visit score - Baseline visit score)
Change from baseline in Meibomian Gland Score (MGS) | 6 weeks
  Meibomian glands on the eyelids assessed by the examiner using a Meibomian Gland Evaluator (MGE) and a slit lamp microscope. An MGE instrument applies a standardized force simulating the pressure of a deliberate blink allowing eye care professionals to observe meibomian gland functionality through a slit lamp. 5 glands in 3 zones (nasal, medial, temporal) evaluated for each eye and scored from 0 to 3, with a resultant overall score (MGS) of 0 to 45 for each eye. Scoring as follows: 0 = no secretion (worst), 1 = inspissated, 2 = cloudy, 3 = clear liquid (best). A higher change from baseline score indicates an improvement in meibomian gland function

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wroblewski, MD, Principal Investigator — George Washington MFA
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No